CLINICAL TRIAL: NCT05805722
Title: Building a Comprehensive Tobacco Cessation Program for Cancer Patients and Survivors: "A Breath of Fresh Air"
Brief Title: Comprehensive Tobacco Cessation for Cancer Patients and Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22-19970; HM20026004 (Other: VCU)
Record Dates: First submitted 2023-03-01; First posted 2023-04-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Use Cessation; Cancer
MeSH Terms: conditions — Tobacco Use Cessation; Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Counseling for Tobacco Cessation (Experimental): Behavioral counseling for tobacco cessation consists of psychoeducation in combination with evidence-based behavior change techniques including stimulus control, self-monitoring, goal-setting, implementation planning, and problem-solving. Specific content topics include the harms of smoking/benefits of quitting, coping with cravings and withdrawal, setting a quit date, managing social influences, and relapse prevention.
  Interventions: Behavioral: Behavioral counseling for tobacco cessation
- Observational Arm (No Intervention): Both the behavioral intervention and pharmacotherapy will be conducted as a routine clinical activities (treatment as usual)-not as research activities

INTERVENTIONS:
Behavioral: Behavioral counseling for tobacco cessation — Participants can choose to receive behavioral counseling in group v. individual format:
  Group Sessions: Participants will be offered the opportunity to attend 6 weekly 60-90 minute sessions Individual Sessions: Participants will be offered the opportunity to attend up to 12 30-45 minute sessions on a schedule mutually agreed upon between interventionist and participant
  Arms: Behavioral Counseling for Tobacco Cessation

SUMMARY:
The purpose of this research study is to learn how best to incorporate tobacco cessation treatment into clinical care for cancer patients, survivors, and caregivers.

DETAILED DESCRIPTION:
The goal of this study is to generate knowledge regarding the feasibility and acceptability of integrating tobacco cessation treatment into clinical care for cancer patients, survivors, and caregivers. The evidence base regarding tobacco treatment is solid: pharmacology (nicotine replacement therapy (and/or), bupropion, or varenicline) in combination with behavioral counseling yields the best results with respect to cessation rates. What remains unclear is how best to offer and implement this comprehensive treatment in the context of a cancer center-especially in a patient population facing social determinants of health that may not be in favor of tobacco cessation. Thus, in this study, the investigators are offering the "gold standard" tobacco treatment and assessing feasibility and acceptability of these procedures in order to inform future efforts to optimize treatment delivery for this unique population and setting. The intervention for this protocol was approved for standard of care use.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with study procedures and availability for the duration of the study
* Have a documented history of cancer of any type, whether active or in remission
* Identify as a current or recently-quit tobacco user

Exclusion Criteria:

* Not a VCUHealth patient
* Non English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Consent rate | At enrollment visit
  The number of individuals who consented to participate compared to the number of individuals approached for study participation.
Feasibility: Barriers to participation | At recruitment visit
  Reasons for refusal will be collected for eligible individuals who do not enroll in the study.
Acceptability: Participant satisfaction | Week 6
  Participant satisfaction ratings will be evaluated utilizing a questionnaire assessing participant satisfaction with the behavioral intervention (if applicable) and/or VCUHS pharmacotherapy management (if applicable) will be administered at each follow-up timepoint.
Acceptability: Participant satisfaction | Week 12
  Participant satisfaction ratings will be evaluated utilizing a questionnaire assessing participant satisfaction with the behavioral intervention (if applicable) and/or VCUHS pharmacotherapy management (if applicable) will be administered at each follow-up timepoint.
Acceptability: Participant satisfaction | Week 24
  Participant satisfaction ratings will be evaluated utilizing a questionnaire assessing participant satisfaction with the behavioral intervention (if applicable) and/or VCUHS pharmacotherapy management (if applicable) will be administered at each follow-up timepoint.
Acceptability: Behavioral counseling attendance | 12 weeks
  Participant attendance at scheduled group or 1:1 behavioral intervention sessions
Acceptability: Nicotine replacement therapy adherence | Week 6
  Self-reported adherence to nicotine replacement therapy and/or varenicline or bupropion will be assessed at each follow-up timepoint. In addition, data re: tobacco cessation medication visits will be extracted from participants' EMR (e.g., number of visits, prescriptions written).
Acceptability: Nicotine replacement therapy adherence | Week 12
  Self-reported adherence to nicotine replacement therapy and/or varenicline or bupropion will be assessed at each follow-up timepoint. In addition, data re: tobacco cessation medication visits will be extracted from participants' EMR (e.g., number of visits, prescriptions written).
Acceptability: Nicotine replacement therapy adherence | Week 24
  Self-reported adherence to nicotine replacement therapy and/or varenicline or bupropion will be assessed at each follow-up timepoint. In addition, data re: tobacco cessation medication visits will be extracted from participants' EMR (e.g., number of visits, prescriptions written).

OTHER OUTCOMES:
Change in tobacco use | Baseline to Week 12
  Self-reported change in number of cigarettes smoked
Change in tobacco use | Baseline to Week 24
  Self-reported change in number of cigarettes smoked

CONTACTS AND LOCATIONS:
Overall Officials: Livingstone Aduse-Poku, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No